CLINICAL TRIAL: NCT01779427
Title: Rehabilitation Research and Training Center for Traumatic Brain Injury Interventions--Attention Intervention Management
Brief Title: Attention Intervention Management
Acronym: AIM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on data from pilot study, the PI and program officer have determined that this study was not feasible.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency); University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H133B090010--03
Record Dates: First submitted 2012-12-10; First posted 2013-01-30 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Brain Injury (TBI); Attention Deficit Hyperactivity Disorder (ADHD); Head Injury; Brain Concussion; Head Injuries, Closed
Keywords: traumatic brain injury (TBI); intracranial edema; brain edema; craniocerebral trauma; head injury; brain hemorrhage, traumatic; subdural hematoma; brain concussion; head injuries, closed; epidural hematoma; extra-axial hemorrhage; cortical contusion; wounds and injuries; disorders of environmental origin; trauma, nervous system; brain injuries; attention deficit hyperactivity disorder (ADHD); attention
MeSH Terms: conditions — Brain Injuries, Traumatic; Attention Deficit Disorder with Hyperactivity; Craniocerebral Trauma; Brain Concussion; Head Injuries, Closed; Brain Edema; Brain Hemorrhage, Traumatic; Hematoma, Subdural; Hematoma, Epidural, Spinal; Brain Contusion; Wounds and Injuries; Disorders of Environmental Origin; Trauma, Nervous System; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIM Intervention (Experimental)
  Interventions: Behavioral: AIM
- Wait List Control (Experimental): Participants are in the Wait List Control group for 10 weeks and then they will participate in the AIM Intervention
  Interventions: Behavioral: AIM

INTERVENTIONS:
Behavioral: AIM — An online, 12 week research study to learn if a computer-based intervention that provides direct attention and metacognitive strategy development can improve attention, memory, and executive control in adolescents with moderate-to-severe TBI who are experiencing attention difficulties post injury.

SUMMARY:
This is a research study to learn if a computer-based intervention that provides direct attention and metacognitive strategy development can improve attention, memory, and executive control in adolescents with moderate-to-severe TBI who are experiencing attention difficulties post injury.

DETAILED DESCRIPTION:
Impairments in attention are among the symptoms most frequently reported by parents and teachers following pediatric traumatic brain injury (TBI_. These cognitive disabilities are responsible for a wide range of academic and adjustment issues. Broadly defined, attention encompasses all of the mental processes, operations, and systems requisite for acquiring and applying information. It interacts with other cognitive functions including perception, memory/learning, organization, and reasoning; attention is core to the integration of those systems. A number of different attentional subcomponents with interconnected neural systems have been identified and shown to be differentially disrupted following trauma and other brain disorders, including maintenance or sustained attention, attentional selectivity, attentional capacity, and ability to effectively shift attention. Given the prevalence of attention difficulties and secondary attention deficit hyperactivity disorder (ADHD) following TBI, it is imperative to identify treatments to effectively address attention impairments.

The study will develop and pilot the Attention Intervention and Management program (AIM). AIM focuses on direct attention training in conjunction with metacognitive strategy training. Strategies are designed to improve focus and self regulation, reduce distractions, and enhance problem solving in academic settings. Integration of attention training and metacognitive strategies will help to ensure that the student can apply the skills across settings and situations.

The Randomized Controlled Trial (RCT) in Phase 2 of this project will address two interrelated hypotheses:

Hypothesis 1: Children receiving the Attention Intervention and Management (AIM) program will evidence better performance on standardized tests of attention and executive functions (EF) than those in the wait list control (WLC) group.

Hypothesis 2: Children receiving AIM will have fewer attention and EF problems than those in the WLC on parent and teacher rating scales of attention and EF.

Participants will include children ages 10-18 with significant evidence of attentional impairments.

ELIGIBILITY:
Inclusion Criteria:

* ages 10-18
* significant evidence of attentional impairments
* moderate to severe TBI
* time since injury at least 6 months
* completion of inpatient rehabilitation (if needed
* English as the primary spoken language in the home.

Exclusion Criteria:

* Child does not live with parents or guardian
* Child or parent has history of hospitalization for psychiatric problem
* TBI is a result of child abuse
* Child suffered a non-blunt injury (e.g., projectile wound, stroke, drowning, or other form of asphyxiation)
* Diagnosed with moderate or severe mental retardation, autism, or a significant developmental disability

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Parent Report Measures | 3 years

SECONDARY OUTCOMES:
Teacher Report Measures | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shari L Wade, PhD, Principal Investigator — Cincinnati Children's Hosiptal Medical Center; McKay M Sohlberg, PhD, Principal Investigator — University of Oregon
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States